CLINICAL TRIAL: NCT04614090
Title: Is Fast Reversal and Early Surgery (Within 24 h) in Patients on Warfarin Medication With Trochanteric Hip Fractures Safe: A Case-control Study
Brief Title: Fast Reversal of Warfarin and Early Surgery in Patients With Trochanteric Hip Fracture A Case-control Study
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Leif Mattisson, Senior Consultant Orthopaedic Surgeon MD.,Ph.D., Karolinska Institutet
Other Study IDs: Leif Mattisson
Record Dates: First submitted 2020-09-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Trochanteric Hip Fractures; Warfarin Medication; Early Surgery
Keywords: Hip fracture; Surgical treatment; Warfarin; Anticoagulation treatment; Intramedullary nailing
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 99 warfarin patients: warfarin patients were operated within 24 h with a cephalomedullary nail due to a trochanteric or subtrochanteric hip fracture. All patients on warfarin were reversed if necessary to INR≤1.5 before surgery using vitamin K and/or four-factor prothrombin complex concentrate (PCC)
- 99 patients without anticoagulants: As a 1:1 ratio control group matched for age, gender and surgical implant. All patients were operated within 24 h with a cephalomedullary nail due to a trochanteric or subtrochanteric hip fracture.

SUMMARY:
A retrospective case-control study. To evaluate if early surgery within 24hours of troch or subtrochanteric hip fractures using intramedullary nailing is safe in patients on warfarin treatment after fast reversal of the warfarin effect

ELIGIBILITY:
Exclusion Criteria:

* Pathological fracture
* Late presentation to the hospital
* Other injuries

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients on warfarin, with low-energi trauma, >60years, mean 86 years Op at Stockholm South General Hospital (södersjukhuset) between (Jan 1,2011 - Dec 31,2014) Follow-up 1 year, all pat op within 24 hours from hospital arrival to the surgery. Operated with Intramedullary nail due to unstable intertrochanteric (OTA/AO 31A2, A3) or Subtrochanteric fracture (OTA/AO 32A,32B,32C).
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Transfusion rates | Pre-surgery
  Hb value (g/dl)
Transfusion rates | Pre-surgery
  Transfusion rate (n)
Transfusion rates | During the surgery
  Hb value (g/dl)
Transfusion rates | During the surgery
  Transfusion rate (n)
Transfusion rates | 2-4 days after the surgery
  Hb value (g/dl)
Transfusion rates | 2-4 days after the surgery
  Transfusion rate (n)
adverse events | Immediately after the surgery
  Number of patients with a myocardial infarction, stroke, pulmonary embolism, deep venous thrombosis, sepsis, pneumonia, urinary tract infection, pressure ulcer, or any adverse events.
mortality | Immediately after the surgery
  The number of deaths
mortality | 30-days after the surgery
  The number of deaths
mortality | 1 year after the surgery
  The number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Leif Mattisson, Principal Investigator — Stockholm South General Hospital
Locations (1):
- Södersjukhuset, Stockholm, Sjukhusbacken 10, Sweden

REFERENCES:
- [Result] Mattisson L, Lapidus LJ, Enocson A. Is fast reversal and early surgery (within 24 h) in patients on warfarin medication with trochanteric hip fractures safe? A case-control study. BMC Musculoskelet Disord. 2018 Jun 26;19(1):203. doi: 10.1186/s12891-018-2126-3. PMID 29945596